CLINICAL TRIAL: NCT04208451
Title: The Effects of One Month Consumption of Standardized Aronia Melanocarpa Extract on Anemia in Patients on Hemodialysis: Focus on Oxidative Stress and Inflammation
Brief Title: The Effects of One Month Consumption of Standardized Aronia Melanocarpa Extract on Anemia in Patients on Hemodialysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All required data are already collected.
Sponsor: University of Kragujevac (Other)
Collaborators: Pharmanova d.o.o., Obrenovac, Serbia (Unknown)
Responsible Party: Principal Investigator, Isidora Milosavljevic, Assistant professor, University of Kragujevac
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Alixir400protect
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Renal Disease; Dialysis; Complications; Anemia
Keywords: hemodialysis; anemia; oxidative stress; inflammation
MeSH Terms: conditions — Kidney Diseases; Anemia; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients on hemodialysis who consumed one month Standardized Aronia Melanocrpa extract
  Interventions: Dietary Supplement: Alixir 400 Protect

INTERVENTIONS:
Dietary Supplement: Alixir 400 Protect — During 30 days all patients take every day 30ml of Alixir 400 protect

SUMMARY:
In this study are included patients on hemodialysis with anemia (levels of Hemoglobin<110). After baseline measurements tha patients take Standardized Aronia melanocarpa extract for one mont and then all measurements were repeated.

DETAILED DESCRIPTION:
1. Patients The study included 30 patients with chronic kidney failure on dialysis treatment at the Center for Nephrology and Dialysis of the Clinical Center Kragujevac. Inclusion criteria were: regular dialysis treatment for more than 3 months, 3 times a week and hemoglobin values lower than 110g / L. Exclusion criteria were: hemoglobin values lower than 80g/L, the use of antioxidant and immunosuppressive therapy, uncontrolled malignancies, proven active bleeding and presence of systemic inflammation or active infection.
2. Ethical approval The research was conducted with respect to the Helsinki Declaration on Medical Research, the approval of the Ethics Committee of the Clinical Center Kragujevac No 01-14-3039. All subjects provided written informed consent before study enrollment.
3. Used plant extract Standardized Aronia extract (SAE) is official product of pharmaceutical company Pharmanova (Belgrade, Serbia); nevertheless, procedure of extraction was done by EU-Chem company (Belgrade, Serbia). This product contains 400mg/30ml of polyphenols, while the recommended daily dosage is 30ml.
4. Blood sampling Patients included in the study consumed standardized Aronia melanocarpa extract (30ml/day) for 30 days. On the day 0, before SAE consumption, blood samples from all patients were collected for hematologic analyzes, inflammation parameters, oxidative stress parameters and antioxidant protection before the dialysis procedure. All mentioned parameters were determined again after consuming the product, ie. on the 30th day of the study.
5. Analytic Procedures Venous blood samples (2 x 4.5ml) were taken before the start of supplementation (zero day) and at the end of supplementation (30th day). Vacuum tubes with sodium citrate were used for blood sampling. The first sample was used for routine hematologic analyzes, the second sample was used for plasma and erythrocyte lysate extraction in order to determinate redox and inflammatory status.
6. Evaluation of Systemic Redox State Plasma samples were used for determination of the levels of the following pro-oxidants: superoxide anion radical (O2-), hydrogen peroxide (H2O2), nitrites (NO2-) and index of lipid peroxidation measured as thiobarbituric acid reactive substances (TBARS), while the parameters of antioxidative defence system, such as activities of superoxide dismutase (SOD) and catalase (CAT) and level of reduced glutathione (GSH) were determined in erythrocytes lysates samples.

   A) Index of lipid peroxidation (TBARS) determination The degree of lipid peroxidation in the plasma samples was estimated by measuring TBARS, using 1% thiobarbituric acid in 0.05 NaOH, which was incubated with the sample at 100°C for 15 min and measured at 530 nm. TBA extract was obtained by combining 0.8 ml sample and 0.4 ml trichloro acetic acid (TCA); afterwards, the samples were put on ice for 10 min and centrifuged for 15 min at 6000 rpm. (1).

   b) Nitrite determination (NO2-)

   Nitric oxide (NO) decomposes rapidly to form stable nitrite/nitrate products. The NO2- level was measured and used as an index of NO production, using Griess's reagent. For NO2 - determination in plasma 0.1 ml 3 N PCA (perchloride acid), 0.4 ml 20 mM ethylenediaminetetraacetic acid (EDTA) and 0.2 ml plasma were put on ice for 15 min, then centrifuged for 15 min at 6000 rpm. After pouring off the supernatant, 220 μl K2CO3 was added. Nitrites were measured at 550 nm. (2)
   1. Superoxide anion radical determination (O2-)

      Superoxide anion radical concentrations in plasma samples were measured using the NTB (Nitro Blue Tetrazolium) reagent in TRIS buffer (assay mixture). The measurement was performed at a wavelength of 530 nm. (3).
   2. Hydrogen peroxide determination (H2O2)

      The measurement of H2O2 was based on the oxidation of phenol red by H2O2 in a reaction catalyzed by horseradish peroxidase. Two hundred microlitres of perfusate or plasma was precipitated using 800 mL of freshly prepared phenol red solution; 10 μL of (1:20) horseradish peroxidase (made immediately before use) was subsequently added. The level of H2O2 was measured at 610 nm (4).
   3. Determination of reduced glutathione (GSH)

      The level of reduced glutathione (GSH) was determined based on GSH oxidation via 5,5-dithiobis-6,2-nitrobenzoic acid. GSH extract was obtained by combining 0.1 ml 0.1% EDTA, 400 μl hemolysate, and 750 μl precipitation solution (containing 1.67 g metaphosphoric acid, 0.2 g EDTA, 30 g NaCl, and filled with distilled water until 100 ml; the solution is stable for 3 weeks at +4C°). The level of GSH was measured at 420 nm (5).
   4. Determination of antioxidant enzymes (SOD, CAT)

   Isolated RBCs were washed three times with three volumes of ice-cold 0.9 mmol/l NaCl, and hemolysates containing about 50 g Hb/l were used for the determination of CAT activity. CAT buffer, prepared hemolysate sample, and 10 mM H2O2 were used for CAT determination. Detection was performed at 360 nm. SOD activity was determined by the epinephrine method. Hemolysate was mixed with carbonate buffer, and then epinephrine was added. Detection was performed at 470 nm (6-10).
7. Evaluation of the inflammatory status In order to evaluate the inflammatory status of patients, following parameters were measured at both points of interest (0 and 30th day): serum C-reactive protein concentration - CRP and tumor necrosis factor concentration - TNF-α.

   The serum C- reactive protein (CRP) concentration was determined by the turbidimetric method on the Olympus AU680. The normal serum CRP concentration is ≤ 5 mg/L. Microinflammation is defined as the concentration of CRP in the serum of 5 mg/L.

   Plasma TNF-α concentrations were determined by enzyme linked immunoadsorbent assay (ELISA) using commercially available high sensitivity indirect sandwich enzyme-linked immunosorbent assay (Sigma Aldrich).
8. Evaluation of the hematological parameters

   At both points of interest, the values of the following haematological parameters in all patients were analyzed:

   Erythrocytes (Er), hemoglobin (Hb), hematocrit (Hct), erythrocyte index- mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), serum lactate dehydrogenase concentration (LDH), serum haptoglobin concentration and iron status: serum iron concentration, ferritin; total iron binding capacity (TIBC), unsaturated iron binding capacity (UIBC), transferrin saturation (TSAT), haptoglobin.
9. Statistical Analysis IBM SPSS Statistics 20.0 Desktop for Windows was used for statistical analysis. Shapiro-Wilk test was used to check the distribution of data. Statistical comparisons were performed using the one-way analysis of variance (ANOVA) tests with a Tukey's post hoc test for multiple comparisons, in the case of normal distribution of data between groups, while Kruskal-Wallis was used for comparison between groups where the distribution of data was different than normal. Values of p < 0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* regular dialysis treatment for more than 3 months, 3 times a week
* hemoglobin values lower than 110g / L

Exclusion Criteria:

* hemoglobin values lower than 80g/L,
* the use of antioxidant and immunosuppressive therapy,
* uncontrolled malignancies,
* proven active bleeding
* presence of systemic inflammation or active infection

Ages: 37 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Anemia control | two months
  The iron levels Unit µmol/l
Anemia control | two months
  The hemoglobin levels Unit g/l
Anemia control | two months
  The ferritin levels Unit ng/ml
Anemia control | two months
  The transferrin levels Unit g/l

SECONDARY OUTCOMES:
Oxidative stress | two months
  Superoxide anion radical, Hydrogen peroxide, Nitrites Units nmol/ml
Oxidative stress | two months
  Superoxide dismutase, Catalase Units U/g Hb x 1000
Oxidative stress | two months
  Reduced glutathione Unit nmol/l RBC x 1000

OTHER OUTCOMES:
Inflammation | two months
  The parameters of inflammation CRP Unit mg/l
Inflammation | two months
  The parameters of inflammation TNF alpha Unit pg/ml
Inflammation | two months
  The parameters of inflammation white blood cells Unit x 1000000000 cells/l

CONTACTS AND LOCATIONS:
Overall Officials: Isidora Milosavljevic, Principal Investigator — Department of pharmacy, University of Kragujevac
Locations (1):
- Faculty of Medical Science, Kragujevac, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milosavljevic I, Jakovljevic V, Petrovic D, Draginic N, Jeremic J, Mitrovic M, Zivkovic V, Srejovic I, Stojic V, Bolevich S, Andjelkovic N. Standardized Aronia melanocarpa extract regulates redox status in patients receiving hemodialysis with anemia. Mol Cell Biochem. 2021 Nov;476(11):4167-4175. doi: 10.1007/s11010-021-04225-y. Epub 2021 Jul 29. PMID 34327604